CLINICAL TRIAL: NCT05405361
Title: A Long-term Extension of the ARGX-117-2002 Trial to Evaluate the Long-term Safety and Tolerability, Efficacy, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of ARGX-117 in Adults With Multifocal Motor Neuropathy
Brief Title: A Clinical Trial to Investigate the Long-term Safety and Tolerability, Efficacy, Pharmacodynamics, Pharmacokinetics, and Immunogenicity of ARGX-117 in Adults With Multifocal Motor Neuropathy
Acronym: ARDA+
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ARGX-117-2003; 2023-507052-69-00 (EU CTIS Number)
Record Dates: First submitted 2022-05-17; First posted 2022-06-06 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Multifocal Motor Neuropathy (MMN)

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: During the double-blinded rollover treatment period (DTP),the investigator, trial nurse/coordinator, participant, and the sponsor's designated contract research organization (CRO), and sponsor trial team (except the sponsor's clinical trial supplies team) are blinded to IMP. The interactive response technology (IRT) system is used for blinding.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARGX-117 (Experimental): Participants receiving ARGX-117 during the double-blinded treatment period (DTP) and the open-label treatment period (OLTP)
  Interventions: Biological: ARGX-117
- Placebo (Experimental): Participants receiving placebo during the double-blinded treatment period (DTP) and receiving ARGX-117 during the open-label treatment period (OLTP)
  Interventions: Biological: ARGX-117; Other: Placebo

INTERVENTIONS:
Biological: ARGX-117 — Intravenous administration of ARGX-117
Other: Placebo — Intravenous administration of placebo
  Arms: Placebo

SUMMARY:
This trial is an extension of the antecedent trial ARGX-117-2002. It is a multicenter trial that has been designed to evaluate the long-term safety and tolerability, efficacy, immunogenicity, Pharmacokinetics (PK), and Pharmacodynamics (PD) of ARGX-117 Intravenously (IV) in adults with Multifocal Motor Neuropathy (MMN). The trial will include a double-blinded rollover treatment period (DTP), an open-label treatment period (OTP), and a safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Capable of providing signed informed consent and complying with protocol requirements. Participants must be able to read and write.
* Must have completed the double-blinded treatment period of the ARGX-117-2002 trial and considered to be eligible for treatment with ARGX-117.

Exclusion Criteria:

* Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection.
* Clinical evidence of other significant serious diseases, have had a recent major surgery, or who have any other condition, in the opinion of the investigator, that could confound the results of the trial or put the participant at undue risk.
* Currently participating in another interventional clinical study.
* Pregnant or lactating or intend to become pregnant during the trial or within 15 months after last dose of the study drug.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety outcomes based on adverse event (AE) monitoring. | Until marketing authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first

SECONDARY OUTCOMES:
Change from baseline in the mMRC-10 sum score | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The modified Medical Research Council (mMRC) sum score evaluates motor strength/weakness from predetermined muscle groups (upper and lower limbs). The higher the score, the better the muscle strength
Proportion of participants showing a deterioration of at least 2 points in mMRC-10 sum score | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The modified Medical Research Council (mMRC) sum score evaluates motor strength/weakness from predetermined muscle groups (upper and lower limbs). The higher the score, the better the muscle strength.
Change from baseline in the mMRC-14 sum score | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The modified Medical Research Council (mMRC) sum score evaluates motor strength/weakness from predetermined muscle groups (upper and lower limbs). The higher the score, the better the muscle strength.
Proportion of participants showing a deterioration of at least 2 points in the mMRC-14 sum score | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The modified Medical Research Council (mMRC) sum score evaluates motor strength/weakness from predetermined muscle groups (upper and lower limbs). The higher the score, the better the muscle strength.
Change from baseline in the average score of the 2 most important muscle groups as assessed by the mMRC-14 sum score | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The modified Medical Research Council (mMRC) sum score evaluates motor strength/weakness from predetermined muscle groups (upper and lower limbs). The higher the score, the better the muscle strength.
Change from baseline in GS | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The grip strength (GS) will be measured by using a Martin-Vigorimeter. Each GS measurement will consist of 3 repeated contractions with the participant's maximal effort. The duration of each contraction will be 3 seconds. 3 repetitions will be executed consecutively by the right hand followed by 3 repetitions of the left hand. There will be a 30-second rest period between each of the 3 repetitions and a 2-minute rest period between each hand.
Proportion of participants with a decline of >30% in GS | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The grip strength (GS) will be measured by using a Martin-Vigorimeter. Each GS measurement will consist of 3 repeated contractions with the participant's maximal effort. The duration of each contraction will be 3 seconds. 3 repetitions will be executed consecutively by the right hand followed by 3 repetitions of the left hand. There will be a 30-second rest period between each of the 3 repetitions and a 2-minute rest period between each hand.
Change from baseline in the MMN-RODS | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The Rasch-Built Overall Disability Scale for MMN (MMN-RODS) is a disease specific patient-reported outcome instrument constructed specifically to capture activity limitations in patients with MMN. The total score varies between 0 (worst outcome) and 50 (best outcome).
Change from baseline in the average time for the upper extremity (arm and hand) function (9-HPT, or timed pegboard test) | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The 9-Hole Peg Test (9-HPT) is a quantitative measure of upper extremity (arm and hand) function. Both the dominant and nondominant hands will be tested twice (2 consecutive trials of the dominant hand, followed immediately by 2 consecutive trials of the nondominant hand).
Proportion of participants by level of severity on each dimension of the EQ-5D-5L | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The Euro-Quality of Life 5 Dimensions 5 Levels (EQ-5D-5L) comprises 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Scores for each dimension include 5 levels: no problem, slight problem, moderate problem, severe problem, and extreme problem.
Change from baseline in EQ-5D-5L visual analog scale (VAS) | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  A vertical visual analog scale (VAS) is included in the EQ-5D-5L. Participants mark their health status from 0 (the worst health you can imagine) to 100 (the best health you can imagine).
Change from baseline in the CAP-PRI | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The Chronic Acquired Polyneuropathy Patient-Reported Index (CAP-PRI) includes the assessment of 15 items. The total score varies between 0 (best outcome) and 30 (worst outcome)
Change from baseline in the 9-item FSS | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  In the 9-item Fatigue Severity Scale (FSS) fatigue levels are rated from 1 to 7. A low value indicates that the statement is not very appropriate whereas a high value indicates agreement.
Values of the PGIC scale | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The Patient Global Impression of Change (PGIC) is a 7-point scale depicting a participant's rating of overall improvement. The lower the score, the better the improvement.
Proportion of participants by level of severity of MMN as assessed by PGIS | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The Patient Global Impression of Severity (PGIS) is a 7-point scale depicting a participant's rating of overall illness severity. Higher scores mean a higher severity.
Values for work-related and household chore activities of the HRPQ | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
  The Health-Related Productivity Questionnaire (HRPQ) provides data related to missed hours at work or educational activities and reduced effectiveness during any attempted work. These criteria form an important portion of work-related productivity and will be used to assess health-related and work-related productivity in the trial.
Serum concentrations for ARGX-117 | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
Change from baseline in free C2, total C2, functional complement activity (CH50). | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first
Incidence of antidrug antibodies (ADA) against ARGX-117 | Until market authorization of ARGX-117, assessed up to 70 months or treatment discontinuation, whichever comes first

CONTACTS AND LOCATIONS:
Locations (27):
- United States (6):
  - HonorHealth Neurology, Scottsdale, Arizona
  - NorthShore University HealthSystem, Glenview, Illinois
  - University of Minnesota, Minneapolis, Minnesota
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvania - Perelman Center for Advanced Medicine, Philadelphia, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
- Medizinische Universitat Wien (Medical University of Vienna), Vienna, Austria
- AZ Sint-Lucas, Ghent, Belgium
- University Health Network, Toronto, Canada
- France (4):
  - CHU Bordeaux - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital Roger Salengro (CHU de Lille), Lille
  - CHU de Nice, Nice
  - Hôpital de la Pitié Salpétrière, Paris
- Germany (2):
  - Universitätsklinikum Essen, Essen
  - Universitatsmedizin Gottingen (UMG) Georg-August-Universitaet, Göttingen
- Italy (4):
  - IRCCS Ospedale San Raffaele S.r.l., Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Azienda Ospedaliera Sant' Andrea, Rome
  - IRCCS Humanitas Research Hospital, Rozzano
- Universitair Medisch Centrum Utrecht, Utrecht, Netherlands
- Poland (2):
  - Michalski i Partnerzy Lekarze Spolka Partnerska, Krakow
  - Warszawski Uniwersytet Medyczny, Warsaw
- Spain (3):
  - Hospital Universitario Vall d'Hebron, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
- United Kingdom (2):
  - Queen Elizabeth University Hospital, Glasgow
  - Oxford University Hospitals NHS Trust, Oxford

IPD SHARING:
Plan to Share IPD: No